CLINICAL TRIAL: NCT02805673
Title: Osteopathic Support Evaluation of Fibromyalgia Patients
Acronym: FMostéo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00687-40
Record Dates: First submitted 2016-01-18; First posted 2016-06-20 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Fibromyalgia
Keywords: Osteopathy; Support; Treatment; Pain; Quality of Life
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Osteopathic Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSTEO group (Experimental): usual medical treatment + 6 osteopathic interventions
  Interventions: Procedure: Osteopathy
- witness group (No Intervention): usual medical treatment

INTERVENTIONS:
Procedure: Osteopathy
  Arms: OSTEO group

SUMMARY:
At present, the literature does not account for much of scientific data on the assessment of osteopathic intervention for patients with (Fibromyalgia) FM. The investigators propose a pilot study evaluating the efficacy of osteopathic care, consists of several osteopathic interventions in the treatment of FM, in order to improve the painful experiences of FM patients. This study must include 44 patients with FM according to (American College of Rheumatology) ACR criteria and followed the University Hospital of Caen.

The osteopathic care will last eight months and will be followed by a report three months after the end of osteopathic interventions. This in order to evaluate the effect in the short term and long term, of osteopathic care in patients with FM.

ELIGIBILITY:
Inclusion Criteria:

* FM patient diagnosed according to the ACR criteria.
* Patient Having realized biological balances excluding any underlying pathology that may be causing the pain.
* Patient Over 18 years followed at Caen University Hospital.
* Patient Treated with drugs to its FM.
* Patient Being informed and having signed his consent.
* Patient Affiliated to the social security system.
* French-Patient.

Exclusion Criteria:

* FM undiagnosed according to the ACR criteria.
* Patient Showing against -indications to the osteopathic surgery.
* Patient Treated by manual therapy ( physiotherapy, osteopathy, acupuncture... ) during the trial and during the three months preceding the study.
* Concomitant Maladie (type cancers, cardiovascular diseases, rheumatic diseases ) or all diseases causing bone pain and myalgia.
* Important Surgery of less than 3 months.
* Inability to submit to medical monitoring study for geographical or social reasons.
* Inclusion The subject in another biomedical research protocol for this study.
* Women Pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for pain | chenge between Day 232 - Day 0

SECONDARY OUTCOMES:
Visual Analogue Scale for pain | change after Week 6, Week 12, Week 18, Week 24, Week 32, Week 38 and day 301, compared to day 0
QDSA score | at day 232 until day 301 and compared to day 0
SF-36 score | at day 232 until day 301 and compared to day 0
number of tender points | at day 232 to day 301 and compared to day 0

CONTACTS AND LOCATIONS:
Overall Officials: Françoise CF COURTHEOUX, MD, Principal Investigator — CHU CAEN
Locations (1):
- CHU Caen, Caen, France